CLINICAL TRIAL: NCT02935296
Title: Integrated Treatment and Prevention for People Who Inject Drugs: A Vanguard Study for a Network-based Randomized HIV Prevention Trial Comparing an Integrated Intervention Including Supported Antiretroviral Therapy to the Standard of Care
Brief Title: Integrated Treatment and Prevention for People Who Inject Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 074; UM1AI068619 (NIH)
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: HIV Positive
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard of Care
- Integrated Intervention (Experimental): Standard of care plus an integrated system of psychosocial counseling and systems navigation for HIV treatment and Substance Use treatment
  Interventions: Behavioral: Integrated Intervention

INTERVENTIONS:
Behavioral: Integrated Intervention — systems navigation, psychosocial counseling
  Arms: Integrated Intervention

SUMMARY:
The purpose of this study is to determine the feasibility of a future trial that will assess whether an integrated intervention combining psychosocial counseling and supported referrals for antiretroviral therapy (ART) at any CD4 cell count and substance use treatment for HIV-infected people who inject drugs (PWID) will reduce HIV transmission to HIV-uninfected injection partners, as compared to routine care dictated by national guidelines for HIV-infected PWID.

DETAILED DESCRIPTION:
This is a multi-site, two-arm, randomized, vanguard study. Network units will consist of an HIV-infected index participant and his/her HIV-uninfected network injection partner(s). Network units will be randomized to the intervention or standard of care arms in a 1:3 ratio, stratified by site. To assess feasibility of the intervention, additional interviews will be conducted with study staff (systems navigators and counselors) and clinic-based stakeholders at each study site.

Approximately 500 Index participants and their partners will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Index participants:

* Age 18-45 years at the Screening visit (age verification procedures will be defined in the Study Specific Procedures [SSP] Manual)
* Able to provide informed consent
* Active injection drug user, defined as self-report of: a) injecting drugs approximately two or more times per week for the past three months, and b) ability to identify the anatomical location of the most recent injection site, as determined by study staff
* Reports sharing needles/syringes or drug solutions at least once in the last month
* HIV-infected based on a study-defined testing algorithm (defined in the SSP Manual)
* Viral load ≥1,000 copies/mL at Screening
* Willing and able to identify, recruit, and have enrolled at least one HIV-uninfected network injection partner who is eligible for study participation according to the criteria below
* Have no plans to move outside the study area for at least one year after study enrollment
* Willing to participate in intervention activities, including regular phone contact

HIV uninfected injection partners:

* Age 18-45 years at the Screening visit (age verification procedures will be defined in the SSP Manual)
* Able to provide informed consent
* Active injection drug user, defined as: a) self-report of injecting drugs approximately two times per week for the past three months, and b) ability to identify the anatomical location of the most recent injection site, as determined by study staff
* Confirmed injection partner, using referral identification cards, of index participant within the past 1 month
* HIV-uninfected based on the study-defined testing algorithm* (defined in the Study SSP Manual)
* Have no plans to move outside the study area for at least one year after study enrollment

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1281 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
HIV incidence among network injection partners of index participants | 18 months
  Number of HIV seroconversions to partners to control arm Index participants
enrollment and retention of HIV-infected PWID and their HIV-uninfected network injection partners | 18 months
  Number of participants enrolled, and number of participants with a final study visit.

SECONDARY OUTCOMES:
HIV incidence among network injection partners of index participants in the intervention arm | 18 months
  Number of HIV seroconversions to partners of Intervention arm participants
Engagement in care for ART treatment services of control arm vs intervention | 18 months
  Number of participants in both arms who report being in ART (case report forms) care, as well as testing stored plasma for HIV RNA suppression
Number of participants in either arm engaged in substance use treatment | 18 months
  self reported on case report forms
size and stability of drug using networks | 18 months
  self reported data via questionnaire of drug sharing habits and partners at each study visit
social harms and benefits | 18 months
  self report via questionnaire
phylogenetics to describe HIV transmission dynamics | 18 months
  stored plasma samples from those persons who are HIV positive and those who become HIV positive during the study

CONTACTS AND LOCATIONS:
Overall Officials: William Miller, MD, Study Chair — Ohio State University
Locations (3):
- CIPTO, Jakarta, Indonesia
- Ukrainian Institute on Public Health Policy, Kiev, Ukraine
- Pho Yen Health Center, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No
no individual data will be shared

REFERENCES:
- [Derived] Sivay MV, Grabowski MK, Zhang Y, Palumbo PJ, Guo X, Piwowar-Manning E, Hamilton EL, Viet Ha T, Antonyak S, Imran D, Go V, Liulchuk M, Djauzi S, Hoffman I, Miller W, Eshleman SH. Phylogenetic Analysis of Human Immunodeficiency Virus from People Who Inject Drugs in Indonesia, Ukraine, and Vietnam: HPTN 074. Clin Infect Dis. 2020 Nov 5;71(8):1836-1846. doi: 10.1093/cid/ciz1081. PMID 31794031
- [Derived] Miller WC, Hoffman IF, Hanscom BS, Ha TV, Dumchev K, Djoerban Z, Rose SM, Latkin CA, Metzger DS, Lancaster KE, Go VF, Dvoriak S, Mollan KR, Reifeis SA, Piwowar-Manning EM, Richardson P, Hudgens MG, Hamilton EL, Sugarman J, Eshleman SH, Susami H, Chu VA, Djauzi S, Kiriazova T, Bui DD, Strathdee SA, Burns DN. A scalable, integrated intervention to engage people who inject drugs in HIV care and medication-assisted treatment (HPTN 074): a randomised, controlled phase 3 feasibility and efficacy study. Lancet. 2018 Sep 1;392(10149):747-759. doi: 10.1016/S0140-6736(18)31487-9. PMID 30191830

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT02935296/Prot_ICF_000.pdf